CLINICAL TRIAL: NCT05854732
Title: Comparison of Uninclined and Inclined Treadmill Training on, Total Body Fat, Lipid Profile and Quality of Life In Obese Adults.
Brief Title: Comparison Of Uninclined And Inclined Treadmill Training In Obese Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01409 FARYAL SHAKOOR
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Obesity
Keywords: Quality of Life; Cholesterol; Exercise; Physical Activity; Lipid Profile; Obesity; Treadmill
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclined Treadmill Training Group (Experimental): The Inclined Treadmill Training Group will be considered as an Experimental group with fixed speed of 5.0 mph and increased inclination of 1% after every one minute. The FITT program for the participants will be:
  * Warmup: 5 mints
  * Frequency: 5days/week for 4 weeks.
  * Intensity: fixed speed of 5.0 mph and increased inclination of 1% after every one minute.
  * Time: 30 minutes
  * Type: 1% Inclined treadmill
  * Cool down: 5 mints
  Interventions: Other: Inclined Treadmill Training
- Uninclined Treadmill Training Group (Active Comparator): The uninclined Treadmill Training Group will be considered as active comparator with no inclination of the treadmill and speed of 5.0 mph. The FIIT program for the participants will be:
  * Warmup: 5 mints
  * Frequency: 5days/week for 4 weeks.
  * Intensity fixed speed of 5.0 mph and no inclination.
  * Time: 30 minutes
  * Type: uninclined treadmill
  * Cool down: 5 mints
  Interventions: Other: Uninclined Treadmill Training

INTERVENTIONS:
Other: Inclined Treadmill Training — Research subjects will be included in the study according to the inclusion criteria and would be randomized into 2 groups, namely inclined treadmill training group and uninclined treadmill training group and will receive intervention for 6 weeks. The participants will be considered as a experimental group with fixed speed of 5.0 mph and increased inclination of 1% after every one minute. FIIT FORMULA will be considered while providing intervention for 5 days per week to the subjects of each group. The FITT program for the participants will be starting with Warmup of 5 mints with Frequency of 5days/week for 6 weeks with fixed speed of 5.0 mph and increased inclination of 1% after every one minute for 30 minutes ending with Cool down for 5 minutes.
  Arms: Inclined Treadmill Training Group
Other: Uninclined Treadmill Training — Research subjects will be included in the study according to the inclusion criteria and would be randomized into 2 groups, namely inclined treadmill training group and uninclined treadmill training group and will receive intervention for 6 weeks. The participants will be considered as a active comparator with fixed speed of 5.0 mph and fixed inclination. FIIT FORMULA will be considered while providing intervention for 5 days per week to the subjects of each group. The FITT program for the participants will be starting with Warmup of 5 mints with Frequency of 5days/week for 6 weeks with fixed speed of 5.0 mph and fixed inclination for 30 minutes ending with Cool down for 5 minutes.
  Arms: Uninclined Treadmill Training Group

SUMMARY:
The goal of this clinical trial is to compare the effects of inclined and uninclined treadmill training on total body fat, lipid profile and quality of life in obese adults. The main question it aims to answer is :

Will there be difference between the effectiveness of inclined and uninclined treadmill training on total body fat, lipid profile and quality of life in obese adults.

Participants will be divided into group A and Group B. Group A participants will be considered as a control group with no inclination of the treadmill and speed of 5.0 mph. Whereas Group B participants will be considered as an interventional group with fixed speed of 5.0 mph and increased inclination of 1% after every one minute.

DETAILED DESCRIPTION:
Obesity is defined as an excessive or abnormal fat accumulation, with body mass index i.e. BMI ≥ 30kg/m2 presenting multiple conditions related to health. Globally which is associated with high rate of mortality and morbidity and low levels of quality of life in adults. Trainings that include moderate and high intensity exercises are believed to be crucial preventive and anti-obesity treatment strategy now a day. Physical activity is a modifiable factor for obesity. Regular physical activity (PA) is an important component of overall well-being of humans and is well known to improve cardiorespiratory fitness, lipid profile, quality of life which are all negatively correlated with the risks of multiple chronic disease. Treadmill exercises are one of the most commonly known exercise therapy models. It can be modified with inclination like 10 degrees which lies in high intensity activity with HR of 80-90%., uninclined treadmill lies in category of moderate intensity physical activity with HR of 55-60%.Advance studies states that HIIT treadmill with variations in inclination is a good way to decrease body fat mass percentage in obese/overweight individuals. In this study Measurements of the anthropometrics of body like bodyweight, BMI (body mass index), WHR (waist and hip ratio), and body fat mass were calculated pre and post the intervention which shows that there was significant decrease in body fat mass percentage according to study.

Literature was reviewed regarding treadmill training effect on total body fat, and lipid profile in different groups of population. The purpose of this study will be to assess the effect of uninclined and inclined treadmill training on obese adults and its effect on calorie burn. This study will help to determine whether which treadmill training is effective to get more benefits on health in less time and on lipid profile and total body fat in obese adults.

ELIGIBILITY:
Inclusion Criteria:

Participants falling in this category would be recruited into the study.

* Males & females
* Body Mass Index (BMI)> 30 kg / m2 (10).
* Age: 18-25
* Physically independent
* Body fat percentage > 25%

Exclusion Criteria:

Participant failing to fall in this category would be excluded of the study.

* Pregnancy
* Nutrition
* Steroid injections in last 6 months
* Psychomotor dysfunction
* Any infection.
* Any neurological and musculoskeletal problems.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Total Body Fat | 6 Weeks
  To estimate the overall amount of body fat, the skinfold thickness is measured using a skinfold caliper. This approach is predicated on the idea that subcutaneous fat is measured by the thickness of the skinfold and that body fat is distributed evenly throughout the body. Four skinfolds are measured in order to determine how much body fat is present overall that includes Biceps muscle fold, Thoracic skinfold, Skinfold on the sub scapula and iliac crest skinfold.
Body Mass Index | 6 Weeks
  A scale or balance is a tool used to determine mass or weight.
Lipid Profile Level (cholesterol and triglycerides) | 6 weeks
  The lipid profile test that is used to check amount of cholesterol and triglycerides in blood.
Quality of Life Questionnaire | 6 Weeks
  The WHOQOL, a tool that measures subjective dimensions of quality of life, was created by the World Health Organization (WHO). One of the most well-known tools for comparing quality of life across cultures is the WHOQOL-BREF, which is accessible in more than 40 languages.Each individual question on the WHOQOL-BREF is graded on a response scale, which is defined as a five-point ordinal scale, with scores ranging from 1 to 5. The scores are then linearly translated to a scale from 0 to 100. The mobility, everyday activities, functional ability, energy, pain, and sleep are all part of the physical health domain that are included in the WHOQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Jawad Naweed, MS-SPT, Principal Investigator — Riphah International University
Locations (1):
- Yusra Medical and Dental College, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No